## **COVER PAGE**

# The Dedicated African American Dad Study NCT number-NCT02412748

Document date- July 7, 2018

**Father Informed Consent Document** 

#### **Father Consent Document**

Investigator: Wrenetha Julion, PhD, MPH, RN

Department Name: Rush University Medical Center College of Nursing Contact Information: 600 S. Paulina, Suite 1055B, Chicago, Il 60612

Telephone Number: (312) 942-6272

Title of Study: The African American Non-resident Fatherhood Program Sponsor: National Institutes of Health/National Institute for Nursing Research

## **©** RUSH

## **Subject Information Sheet and Consent Form**

#### Introduction

This form provides you with information so you can understand the possible risks and benefits of participating in this study; so that you can decide whether or not you want to be a part of this research study. Before deciding whether to participate in this study, you should read the information provided on this document and ask questions regarding this study. Once the study has been explained and you have had all your questions answered to your satisfaction, you will be asked to sign this form if you wish to participate.

#### Why are you invited to participate in this study?

Thank you for your interest in the D.A.A.D. Study. You are being asked to take part in this study because you are an African American father of a young child who you do not live with on a full-time basis. Research studies include only people who choose to take part. Please take your time to make your decision and discuss it with your friends, family and/or physician. Remember that your participation is completely voluntary. There is no penalty if you decide not to take part in this study or decide later that you want to stop participating in this research study. Your care at Rush University Medical Center will not be affected if you decide not to participate.

## What is the purpose of this study?

The purpose of this study is to test out two programs for helping fathers of young children improve their skills taking care of their children. As part of this study you will meet in groups with about 10-12 other fathers over 12 weeks. During that time there will be 9 meetings and 3 scheduled break-weeks, and a booster session that will be scheduled 6 weeks after the groups end.

## How many study subjects are expected to take part in the study?

We plan to have about 180 fathers and 180 mothers take part in this study and all of the fathers and mothers will be signed-up to participate by investigators from Rush. This is currently the only site for this study.

## What will you be asked to do?

If you wish to be a part of this study:

1. You will have to be randomized to participate in either the Fatherhood program called Building Bridges to Fatherhood (BBTF) or the Finance Program called Money Smart (MS). This means that half of the fathers who sign up will participate in BBTF and the

Template Version Date: 8/6/2014

Consent Version Date: 4/19/2016 1 of 6

ORA: 14022704-IRB01-CR03 Date IRB Approved: 7/6/2017 Expiration Date: 7/6/2018

other half will participate in the MS program. Randomization means that the group you participate in will be decided by chance alone (like flipping a coin). Neither you nor the research team members can choose what group you will be in. You will have a one in two chance of being placed in either group. After you are officially signed up for the program, you will be told which group you will participate in.

- 2. Read and sign the "consent form." By signing the consent form you are letting us know that you have read about our project, understand that it is a research study, have had your questions answer, and that you agree to participate in this study. You will be given a copy of this form to keep.
- 3. Complete an interview with a member of the study team at the beginning, middle and end of the study. It will take about 60 minutes to complete this form.
- 4. Meet in groups with about 10-12 other fathers over 12 weeks. During that time there will be 9 meetings, 3 scheduled break-weeks, and a booster session that will be scheduled 6 weeks after the groups end. Each meeting will last for about 2 hours. During these skill-building meetings you will learn information that can help in your role as a father. You will receive free dinner during the group meetings. We will call you to let you know when and where the groups will meet.
- 5. Be willing to have your child's mother or primary caregiver consent to be a part of the study by completing the Child Information Interview and allowing the child to spend time with you. This is very important because we want to get information about the child from both the mother/primary caregiver and the father, when parents don't live together and we want you to have a good relationship with your child. If you decide to stop being a part of this study before it ends, your child's mother/primary caregiver can still give us information about your child. If your child's mother/primary caregiver decides to stop being a part of this study before it ends, you can still be a part of the groups and give us information about your relationship with your child.
- 6. Participate in the group meetings that will be tape recorded to make sure our group leaders are following the guidelines on how the groups should be run. The tape recordings will be destroyed after the project has ended. After you and your child's mother/primary caregiver sign the consent form and complete the interview, your participation in one of the 2 groups will begin.

#### How long will you be in the study?

Altogether you will be participating in the study for about 9 months.

## What are the possible risks of the study?

There is a risk that if you and your child's mother increase your contact with each other that there may be increased conflict between you and her. If this happens, we have a team of 3 professionals (clinical psychologist, mental health nurse specialist and African American male social worker) who you can talk to; and who can help you connect with local community-based resources to get help with solving problems with your child's mother. If you would like more information on these services please contact Dr. Wrenetha Julion, the nurse in charge of this study. There will be no costs related to meeting with members of the study research team, however you will be responsible for any costs related to seeking counseling or obtaining help problem-solving with your child's mother.

This project has been approved by the Rush University Medical Center's Institutional Review Board (IRB). The IRB is a special committee that reviews human research to check that the rules and regulations are followed. We have been meeting with groups of non-resident fathers to help

Template Version Date: 8/6/2014

them stay connected with their children for over 10 years and we have received very positive comments from the fathers who participated in the groups. If any additional risks to participation become known or if new information comes out that may affect your desire to stay in the study, we will let you know in a timely manner. If for any reason this project and, thus your participation is stopped, we will also let you know.

## Are there benefits to taking part in the study?

There may be no direct benefit to you for being in this study, other than the benefit you receive from learning new skills with a group of fathers like yourself. This program could help you and other fathers stay involved in the lives of your children and could help improve your relationship with your child's mother.

## What other options are there?

Other than being a part of another fatherhood group through another agency or in the community, there is no alternative program being offered at this time. If you choose not to participate in the D.A.A.D. study, community group programs would still be available to you. Everyone who is a part of this study has the right to withdraw from the study at any time. Please contact Dr. Wrenetha Julion at 312-942-6272 if you would like to stop participating in the study. We will keep and analyze the data that we have already collected from you. This data will be analyzed without making your identity known.

#### What about confidentiality of your information?

Records of participation in this research project will be maintained and kept confidential as required by law. We will use a code number on all of your questionnaires. Other than this code number, there is no way your answers to the questions can be connected to you. Your answers to questions will be entered into a computer and looked at as part of a group of fathers (180 total). If the results of this project are published, your identity will not be made known. People who are in charge of the agency who gave us the money for this study (NINR), and The Rush Institutional Review Board (IRB) may ask to see the research to make sure that it is being done correctly and ethically, but this will be done without any loss of confidentiality. After five years, the information you have provided to us will have all identifying information removed from it and the records that link the information to you will all be destroyed. The data will then be kept indefinitely until it is determined that they can serve no further useful purposes.

To further protect the confidentiality of your data, we have obtained a Certificate of Confidentiality from the Department of Health and Human Services (DHHS). With this certificate, we cannot be forced (for example by court subpoena) to disclose research information that may identify you in any Federal, State, or local civil, criminal, administrative, legislative, or other proceedings. Disclosure will be necessary, however upon request of federal agencies for audit or program evaluation purposes.

You should understand that a Confidentiality Certificate does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this study. If you give your consent to a third party to receive research information, then we may not use the Certificate of Confidentiality to withhold this information. This means that you and your family must also actively protect your own privacy and the confidentiality of your data.

Finally you should understand that we are not prevented from taking steps including making reports to authorities to prevent serious harm to yourself or others. All members of the

Template Version Date: 8/6/2014

research team are required by law to report child abuse or neglect to the Department of Children and Family Services. In addition, if members of the research team have reason to believe that there is a threat of violence to you or others, we will also report that information to the appropriate authorities.

Confidentiality and disclosure of your personal information is further described in the attachment to this form. The attachment is entitled HIPAA Authorization to Share Personal Health Information in Research (2 pages).

## What are the costs of your participation?

If you choose to participate in the D.A.A.D. Study, there are no additional costs to you other than the cost of your time.

## What financial disclosure(s) apply to this study?

Research studies like this one are designed to determine whether the program affects father involvement in pre-school children. Rush University owns the patent on the program called Building Bridges to Fatherhood (BBTF) being studied. If research shows the program is effective, Rush University would receive profits from any sales and or licensing of the program.

It was determined that the additional payments to Rush were considered unlikely to affect your safety and/or the scientific quality of the study. This recommendation was given to the IRB for its review and approval of this study. If you would like more information, please ask Dr. Julion.

#### Will you be paid for your time?

You will get \$50 every time you complete the interview about you and your child (\$150 total), as compensation for the time you spend being interviewed. In addition, you will be paid \$15 every time you attend each group meeting.

## What happens if you experience a research related injury?

If you experience any injury or illness as a direct result of your participation in this research study, immediate treatment will be provided. However, the cost of that treatment will be billed to you or your insurance company. We do not expect that you will experience any injuries as a result of being in the study. However, Rush University Medical Center has no program for financial compensation or other forms of compensation for injuries which you may incur as a result of participation in this study.

## Whom do you call if you have questions or problems?

Questions are encouraged. If you have any concerns about this or anything else related to this project, or if you experience a research related injury, please call Dr. Wrenetha Julion, who is in charge of this project at (312) 942-6272. You may also choose to get out of this project at any time by calling Dr. Julion at (312) 942-6272. Dr. Julion is a teacher and nurse who works at Rush University Medical Center. If you have any questions about the rights of people who are a part of research studies at Rush please call the Rush Research and Clinical Trials Administration Office at 1-800-876-0722.

#### **Future Research**

There may be other studies that come up in the future that are of interest to you. By checking, the box below, you are agreeing that we may contact you to see if you are eligible and willing to participate in future research. There is no penalty for deciding not to participate.

Template Version Date: 8/6/2014

Consent Version Date: 4/19/2016 4 of 6

| | red in being contacted for future resenterested in being contacted for futur | |
|---|---|---|
| information given or someone ha | | pportunity to ask questions, |
| Name of Subject | Signature of Subject | Date of Signature |
| I attest that all the elements of in | formed consent described in this corterms with the subject. I further attembest of my knowledge. | nsent document have been |
| Signature of Individual Obtaining | _ | Date of Signature |
| document and can attest, to the b<br>the subject or the subject's legali | Obtaining Consent observed the signost of their knowledge, the person sily authorized representative and the this box, the Individual Obtaining (e (below). | igning the consent form is<br>person signing the form has |
| | TRANSLATOR | |
| | nsent document and attest that, to the is the subject or the subject's legally has done so voluntarily. | |
| Signature of Witness/Translator<br>Check here if a separate witness | signature is not necessary. | Date of Signature |
| SIGNATURE OF THE PRINC<br>I attest that I am aware of the enr | CIPAL INVESTIGATOR rollment of this subject in the study of | discussed in this consent |

ORA: 14022704-IRB01-CR03 Date IRB Approved: 7/6/2017 Expiration Date: 7/6/2018

document.

5 of 6

Template Version Date: 8/6/2014

Consent Version Date: 4/19/2016

Signature of the Principal Investigator

Check here if Principal Investigator obtained consent and a separate signature is not required.

ORA: 14022704-IRB01-CR03 Date IRB Approved: 7/6/2017 Expiration Date: 7/6/2018

Template Version Date: 8/6/2014